CLINICAL TRIAL: NCT04569487
Title: Identification of Relevant Biological, Imaging, Mobility and Clinical Markers for Clinical Research in Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DEMAIN
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, cohort study with 2 parallel groups (sarcopenic versus non-sarcopenic population)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenic population (Active Comparator): Diagnosed sarcopenia following definition of the EWGSOP2:
  * Muscle strength assessed by the handgrip test <27 kg
  * Skeletal muscle mass index (Appendicular lean muscle mass) assessed by DXA <7.0 kg/m2
  Interventions: Procedure: Biopsy
- Non sarcopenic population (Active Comparator): Non-sarcopenic population adapted from the EWGSOP2:
  * Muscle strength assessed by the handgrip test ≥ 27 kg
  * Skeletal muscle mass index (Appendicular lean muscle mass) assessed by DXA ≥ 7.0 kg/m2
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Muscle biopsy from vastus lateralis (100-200 mg from non-dominant leg)

SUMMARY:
The objective of this trial is to constitute a cohort of sarcopenic versus non-sarcopenic patients to validate the most relevant biological, imaging, mobility and clinical markers considered individually or in association for the diagnosis of sarcopenic patients.

DETAILED DESCRIPTION:
This trial is part of a Research Program partly funded by a grant from the Walloon region entitled "Development of Markers of Sarcopenia Using an Integrated Approach : From Cell to Human".

Consistent with the above-mentioned observation, there is not only one biological marker that perfectly matches the sarcopenia criteria but there is a range of complementary biomarkers - including but not limited to inflammation markers, products of oxidative damage, serum creatinine and urinary creatinine excretion, endocrine function, urine proteomics panel, N-terminal procollagen peptides, myostatin and agrin fragment - that will together constitute the ideal panel of markers (Fougère et al, 2015). These current biomarkers and the thresholds for correlation with clinical outcomes have to be deeply evaluated in clinical trials before being considered as good biomarkers.

In addition, one research priority is to investigate and define novel biomarkers allowing an improved assessment, characterization and follow-up of elderly people with sarcopenia. Biomarkers derived from blood can indeed easily be measured in a standardized and low-cost way and are therefore very attractive.

This clinical trial aims at confirming the relevance of new soluble markers and validating the most relevant biological (previously and newly identified), imaging, mobility and clinical markers for clinical research in sarcopenia.

Newly identified soluble markers of sarcopenia coming from DEMAIN Research program and using secretomic approach (to be identified in secretome of human myotubes during the program research) using immunoassays on biological fluids.

ELIGIBILITY:
Inclusion Criteria:

Participants will have the following inclusion criteria:

* Male with age ≥ 65 years
* Body Mass Index: 20 < BMI < 35 kg/m2
* Able to understand and having signed an informed consent
* Able to follow the trial procedures

Sarcopenic population: diagnosed sarcopenia following definition of the EWGSOP2:

* Muscle strength assessed by the handgrip test <27 kg for male
* Skeletal muscle mass index (Appendicular lean muscle mass) assessed by DXA <7.0 kg/m2

Non-sarcopenic population: adapted from the EWGSOP2:

* Muscle strength assessed by the handgrip test ≥ 27 kg
* Skeletal muscle mass index (Appendicular lean muscle mass) assessed by DXA ≥ 7.0 kg/m2

Exclusion Criteria:

Participants will have the following exclusion criteria:

* Any clinically significant levels of the safety parameters (Creatine Kinase (CK), activated Partial Thromboplastin Time (aPTT), Prothrombin Time and International Normalized Ratio (PT/INR))
* Any severe, uncontrolled and limiting diseases (e.g. systemic inflammation, infectious diseases, active cancer, neurodegenerative disorders, diabetes) left to the investigator's discretion
* Bed resting for more than 10 days during the 3 months preceding the recruitment
* Immobilization of the lower limb, lasting more than one week during the 3 months preceding recruitment
* Medical treatment with anticoagulant, insulin, immunosuppressant, long-term corticosteroid (over 7.5 mg prednisone or its equivalent)
* Severe incapacity (class IV Steinbrocker Functional Classification - Appendix 2)
* Any treatment that may affect physical performance, muscle function, disrupts study measures or impairs the understanding of consent
* Known acute or severe renal insufficiency (glomerular filtration rate < 30 mL/min/1.73m2)
* Cushing' syndrome
* Known cachexia
* Currently participating or having participated in another therapeutic clinical trial in the three previous months
* Under guardianship or judicial protection

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Identified soluble markers of sarcopenia | 3 months after biopsy
  immunoassays on biological fluids by secretomic approach

SECONDARY OUTCOMES:
Identified imaging marker | within 15 days after Day 0 (baseline visit)
  Appendicular lean muscle mass and adiposity (if possible) using Dual Energy Xray Absorptiometry (DXA)
Determine thePhysical performance | Day 0 (baseline visit)
  Patients realize some physical tests: Short Physical Performance Battery (SPPB that are three physical tests: gait speed, balance test, chair stand test)
Determine the falls risk | Day 0 (baseline visit)
  A global score will be calculated in function of the answers of a Self-administered questionnaire: Morse Fall Scale (MFS; falls risks for elderly)
Identified clinical marker | Day 0 (baseline visit)
  A global score will be calculated in function of the answers of a Self-administered questionnaire: SARC-F
Determine the muscle strength | Day 0 (baseline visit)
  Handgrip muscular strength test (upper body skeletal muscle function) using a hand dynamometer
Evaluate the quality of life | Day 0 (baseline visit)
  A global score will be calculated in function of the answers of a Self-administered questionnaire (SF-36). The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Determine cognitive performance | Day 0 (baseline visit)
  A global score will be calculated in function of the answers of a Self-administered questionnaire: Montreal Cognitive Assessment (MoCA)
Determine the nutrition status | Day 0(baseline visit)
  A global score will be calculated in function of the on Global Leadership Initiative on Malnutrition (GLIM) criteria (Cederholm et al, 2018)
Evaluate the tolerance | 3 months (baseline visit to biopsy)
  Number of Adverse events (AE or Adverse Device Effect or Device Deficiency; will be coded in terms of System Organ Class (SOC) and Low Level Terms (LLT) using the last version of MedDRA) and drop offs

CONTACTS AND LOCATIONS:
Overall Officials: Yves Henrotin, Prof, Study Director — Artialis
Locations (2):
- Belgium (2):
  - Erasme Hospital, Brussels
  - Universitair Ziekenhuis Brussel, Brussels

IPD SHARING:
Plan to Share IPD: No